CLINICAL TRIAL: NCT02282982
Title: Prospective, Multi-Center, Observational Program to Assess RSV Hospitalization Rate in Population of Children at High-risk of Serious RSV Illness Who Received Palivizumab Immunoprophylaxis in Routine Clinical Setting in the Russian Federation
Brief Title: Observational Program to Assess Respiratory Syncytial Virus (RSV) Hospitalization Rate in Population of Children at High-risk of Serious RSV Illness Who Received Palivizumab Immunoprophylaxis
Acronym: SUNRISE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-579
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Immunoprophylaxis; Palivizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants at high-risk of serious RSV illness: Infants who received immunoprophylaxis during the RSV season

SUMMARY:
This was a non-interventional, prospective, multi-center study with no control group designed to assess the effectiveness of palivizumab in a population of infants at high-risk of serious Respiratory Syncytial Virus (RSV) illness (infants born ≤ 35 weeks of gestation and infants ≤24 months with Bronchopulmonary Dysplasia (BPD) or Congenital Heart Disease (CHD)). Participants received immunoprophylaxis during the RSV season, defined as October 2014 through April 2015, in routine clinical settings throughout the Russian Federation.

DETAILED DESCRIPTION:
Participants received intramuscular injections of palivizumab according to physicians' prescription and the local label. The local label recommended 1 month injection intervals between 5 sequential injections at a dose of 15 mg/kg. Participants could have received from 3 to 5 monthly injections of palivizumab during the 2014 - 2015 RSV season and the duration of this study.

ELIGIBILITY:
Inclusion Criteria:

* Planned prescription of palivizumab for immunoprophylaxis during RSV season or participants for whom palivizumab was prescribed and who received the first dose of palivizumab no later than 60 days before enrollment in the study
* Infants at high risk of severe RSV infection defined as fulfilling at least one of the following:

  * Infants born ≤35 weeks gestational age AND are ≤6 months of age at the onset of the RSV season;
  * Infants ≤24 months of age AND with a diagnosis of BPD (defined as oxygen requirement at a corrected gestational age of 36 weeks);
  * Infants ≤24 months of age with hemodynamically significant CHD, unoperated or partially corrected.
* Written authorization to use individual data signed by parents or child representative

Exclusion Criteria:

* Major congenital malformation aside from CHD
* Chronic pulmonary disease other than BPD
* Acute period of any infection
* Contraindication to palivizumab prescription according to local label
* Administration of a product possibly containing RSV-neutralizing antibody within 30 days prior to enrollment or current administration (includes, but is not restricted to, the following: RSV hyperimmunoglobulin, polyclonal intravenous immunoglobulin, cytomegalovirus hyperimmunoglobulin, varicella zoster hyperimmunoglobulin)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants at high-risk of serious Respiratory Syncytial Virus (RSV) illness (infants born ≤ 35 weeks of gestation and infants ≤24 months with Bronchopulmonary Dysplasia (BPD) or Congenital Heart Disease (CHD)) who received immunoprophylaxis during the RSV season defined as October 2014 through April 2015 in routine clinical settings in the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Strugovschikov, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infants at High-risk of Serious RSV Illness
Started | 359
Attended Visit 1 | 359
Attended Visit 2 | 341
Attended Visit 3 | 298
Attended Visit 4 | 194
Attended Visit 5 | 83
Attended Follow-up Visit | 349
Completed | 153
Not Completed | 206
Not completed — Lost to Follow-up | 15
Not completed — Withdrew consent | 2
Not completed — Death | 4
Not completed — Lack of product | 156
Not completed — Palivizumab is ended | 11
Not completed — Other, not specified | 18

BASELINE CHARACTERISTICS:
Population: Infants who received immunoprophylaxis during the RSV season
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 359
Age, Continuous [Mean (Standard Deviation); unit: months] | 3.4 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179
  Male | 180

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Infants Hospitalized for Lower Respiratory Tract Infection (LRTI) With a Positive Respiratory Syncytial Virus (RSV) Diagnostic Test
Description: Hospitalizations for LRTI with positive RSV diagnostic tests were documented at study visits.
Time Frame: Approximately 7 months
Population: Infants who received immunoprophylaxis during the RSV season
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 359
participants | 1

2. Primary Outcome: Proportion of Infants Who Died From a Confirmed Respiratory Syncytial Virus (RSV) Infection
Description: Deaths caused by RSV during the study were to be confirmed by autopsy or clinical history and positive virologic diagnostic tests.
Time Frame: Approximately 7 months
Population: Infants who received immunoprophylaxis during the RSV season
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 359
participants | 0

3. Secondary Outcome: Median Length of Stay (LOS) of Lower Respiratory Tract Infection (LRTI) Hospitalization With a Positive Respiratory Syncytial Virus (RSV) Test
Description: The duration of hospitalizations due to LRTI which were accompanied by a positive RSV diagnostic test was documented.
Time Frame: Approximately 7 months
Population: Participants who were hospitalized due to Lower Respiratory Tract Infection and who had a positive Respiratory Syncytial Virus laboratory diagnostic test
Measure: Median (Full Range); unit: days
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
days | 46 [NA to NA] — Only 1 participant was analyzed for this outcome.

4. Secondary Outcome: Proportion of Participants With Intensive Care Unit (ICU) Admission Among Hospitalized Participants
Description: The number of hospitalized participants admitted to the Intensive Care Unit was documented.
Time Frame: Approximately 7 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
participants | 1

5. Secondary Outcome: Median Length of Stay (LOS) of Participants in the Intensive Care Unit (ICU)
Description: The median length of stay of hospitalized participants in the Intensive Care Unit was calculated.
Time Frame: Approximately 7 months
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
days | 35 [NA to NA] — Only 1 participant was analyzed for this outcome.

6. Secondary Outcome: Proportion of Participants Who Received Supplemental Oxygen While Hospitalized
Description: The proportion of participants who received supplemental oxygen while hospitalized was documented.
Time Frame: Approximately 7 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
participants | 1

7. Secondary Outcome: Proportion of Participants Who Received Mechanical Ventilation While Hospitalized
Description: The proportion of participants who received mechanical ventilation while hospitalized was documented.
Time Frame: Approximately 7 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
participants | 0

8. Secondary Outcome: Proportion of Participants With Missed Doses of Palivizumab
Description: The proportion of participants with missed or delayed doses of palivizumab was documented.
Time Frame: Approximately 7 months
Population: Infants who received immunoprophylaxis during the RSV season
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 359
participants
  1 missed or delayed injection | 61
  2 or more missed or delayed injections | 20

9. Secondary Outcome: Proportion of Participants With Co-morbidities During Hospitalizations
Description: The proportion of participants with co-morbidities during hospitalizations was documented. Co-morbidities were defined by the International Statistical Classification of Diseases 10 revision (ICD-10).
Time Frame: Approximately 7 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
participants | 1

10. Secondary Outcome: Median Duration of Mechanical Ventilation Administration During Hospitalizations
Description: The median duration of mechanical ventilation administration during hospitalizations was calculated.
Time Frame: Approximately 7 months
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
days | 0 [NA to NA] — Only 1 participant was analyzed for this outcome.

11. Secondary Outcome: Median Duration of Oxygen Administration During Hospitalizations
Description: The median duration of mechanical oxygen administration during hospitalizations was calculated.
Time Frame: Approximately 7 months
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 1
days | 30 [NA to NA] — Only 1 participant was analyzed for this outcome.

12. Secondary Outcome: Proportion of Participants With a Particular Co-morbidity
Description: The proportion of participants with co-morbidities was documented. Co-morbidities were defined by the International Statistical Classification of Diseases 10 revision (ICD-10).
Time Frame: Approximately 7 months
Population: Infants who received immunoprophylaxis during the RSV season
Measure: Number; unit: participants
Arm/Group | Infants at High-risk of Serious RSV Illness
Number analyzed (Participants) | 359
participants
  History of bronchopulmonary dysplasia | 148
  History of congenital heart disease | 45

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time of the first dose of palivizumab until the last dose, up to 17 weeks.
Description: Serious adverse events were collected from the time of informed consent until 30 days following the last dose of palivizumab, up to 21 weeks.
Arm/Group | Infants at High-risk of Serious RSV Illness
Serious Adverse Events (participants affected / at risk) | 17/359
Other Adverse Events (participants affected / at risk) | 0/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infants at High-risk of Serious RSV Illness (N=359)
Respiratory tract infection viral (Infections and infestations) | 6
Bronchitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 5
Bronchopneumonia (Infections and infestations) | 2
Otitis media acute (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Ascites (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1
Brain oedema (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Periventricular leukomalacia (Nervous system disorders) | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.